CLINICAL TRIAL: NCT05192317
Title: A Randomized, Parallel Group, Placebo-controlled, Double Blinded Clinical Trial to Evaluate the Efficacy and Safety of the Substance-based Medical Device (Sollievo Fisiolax) in the Treatment of Chronic Constipation.
Brief Title: Administration of a Natural Molecular Complex in Functional Chronic Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: JSB Solutions S.R.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABO-SOLDM-02/21
Record Dates: First submitted 2021-10-22; First posted 2022-01-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Chronic Constipation
Keywords: Chronic Constipation; Medical Device; Sollievo Fisiolax; Natural Molecular Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Sollievo Fisiolax (Experimental): Sollievo Fisiolax
  Interventions: Device: Sollievo Fisiolax
- Arm Placebo (Placebo Comparator): Placebo
  Interventions: Other: Sollievo Fisiolax Placebo

INTERVENTIONS:
Device: Sollievo Fisiolax — Class IIb Medical Device
  Arms: Arm Sollievo Fisiolax
Other: Sollievo Fisiolax Placebo — Placebo
  Arms: Arm Placebo

SUMMARY:
This is a multi-center, randomized, double-blinded placebo controlled trial to evaluate the efficacy and safety of the substance-based medical device (Sollievo Fisiolax) in the treatment of Chronic Constipation.

Treatment period for each patient is 28 days.

DETAILED DESCRIPTION:
According to the criteria of Rome IV, 86 patients diagnosed from chronic constipation will be enrolled by up to ten centers.

The study includes 2 visits at the site center and 1 by phone call.

V-1 (eligibility assessment / screening visit):

* Collection of written informed consent
* Physical examination, including measurement of anthropometric parameters and vital signs (height, weight, diastolic / systolic pressure, heart rate)
* Diagnosis according to Rome IV criteria of chronic functional constipation
* Blood tests: glycemia, creatinine, complete blood count with formula, ALT, AST, ALP, calcium, potassium, sodium, C reactive protein, total bilirubin. Urinalysis.
* Performing a colonoscopy for patients aged> 50 who have not had one performed in the last 5 years.
* Guideline for daily diary to collect the number and the consistency of the evacuations, and whether or not they occur with effort
* Recording of adverse events and concomitant therapies

V0 (confirmation of possession of selection criteria):

* Physical examination, including measurement of anthropometric parameters and vital signs (height, weight, diastolic / systolic pressure, heart rate)
* Randomization 1:1 to Sollievo Fisiolax or Placebo
* Blood and fecal sample collection for the evaluations of the exploratory objectives
* Compliance of the daily diary
* Administration of questionnaires: Gastrointestinal Quality of Life Index (GIQLI), PAC-SYM
* Any changes in concomitant therapies and any adverse events will be recorded.

V1 (end of treatment or discontinuation before study / treatment time; 4 weeks after V0):

* Physical examination, including measurement of anthropometric parameters and vital signs (height, weight, diastolic / systolic pressure, heart rate)
* Returned the Investigational product
* Blood and fecal sample collection for the evaluations of the exploratory objectives.
* Blood tests: glycemia, creatinine, complete blood count with formula, ALT, AST, ALP, calcium, potassium, sodium, C reactive protein, total bilirubin. Urinalysis.
* Blood sampling for the screening of HIV, HCV, HBV and TPHA
* Check of daily diary
* Administration of questionnaires: Gastrointestinal Quality of Life Index (GIQLI), PAC-SYM
* Any changes in concomitant therapies and any adverse events will be recorded

ELIGIBILITY:
Inclusion Criteria:

1. Patient giving written informed consent to participate in the study.
2. Patient of both sexes aged between 18 and 70 years (inclusive)
3. Patient affected by chronic functional constipation according to the Rome IV criteria
4. In patients over the age of 50, negative colonoscopy, i.e. absence of clinically relevant alterations or in any case of critical condition for study participation, performed during the run-in period unless:

at least negative colonoscopy performed in the previous 5 years the symptoms have remained unchanged, if present, from the time of the execution of the (or last, if more than one) colonoscopy

Exclusion Criteria:

1. Hypersensitivity or Suspected or known allergy to one of the components of the products under study
2. Have previously taken the study product
3. Therapy with antibiotics within 4 weeks prior to the screening visit (i.e, prior to the visit V -1)
4. Therapy within 2 weeks of the run-in (i.e., prior to the visit V0) with: Laxatives / fecal softeners / intestinal bulking products; Drugs indicated for the treatment of obesity; probiotics or prebiotics
5. Chronic inflammatory bowel diseases
6. Intestinal diseases of infectious, actinic, endocrine or pharmacologic origin (microscopic colitis)
7. Patients undergoing gastro-intestinal resection
8. Renal, hepatic, haematological, cardiovascular, pulmonary, neurological, psychiatric, immunological, endocrine diseases, if they are clinically significant
9. Patients with malignant neoplasm of any type, or history of malignancy, with the exclusion of patients with a history of extra-intestinal malignant neoplasm surgically removed and no evidence of recurrence within the five years prior to participation
10. Abuse of alcohol, narcotics or psychotropic drugs that can change vigilance and physical perception
11. Presence of a dementia of any type or other possible causes of progressive deterioration of the capacity to understand and of want or psycho-physical disability that reduces the ability to assume as expected the study treatment
12. Obesity (BMI ≥ 30)
13. No adequate reliability or conditions that may lead to a non-compliance / adherence of the patient to the protocol
14. Previous participation in a clinical trial in the last 30 days
15. Patients who for any reason do not agree to guarantee the commitment to keep their diet stable for the study period

    * During the run-in period, in case of severe symptoms, the use of an evacuant to be applied rectally, indicated in constipation and identified by the Investigator, can be used as a "rescue" therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the number of spontaneous complete bowel movement | 28 days
  Response rate (RR) to study treatment, defined by an increase of at least 1 spontaneous complete bowel movement, (SCBM) / weekly from baseline, in at least 75% of the weeks of the treatment period

SECONDARY OUTCOMES:
Patient satisfaction | 7 days, 14 days, 21 days, 28 days
  Composite rate of satisfaction with the treatment and improvement of the symptom complex, with "satisfaction" and "improvement" defined respectively by:
  * a ˃4 score on the following 7-point Likert scale of "satisfaction with treatment":
    1. = extremely dissatisfied,
    2. = very dissatisfied,
    3. = dissatisfied,
    4. = partially satisfied,
    5. = satisfied,
    6. = very satisfied,
    7. = extremely satisfied
  * a score ≥2 on a global change rating scale (-7 to +7: -7 = extremely worsened, 0 = unchanged, +7 = extremely improved).
Change in Stool frequency | through study completion, an average of 1 month
  Post treatment stool frequency increase respect to the Baseline
Change in Patient Assessment of Constipation-Symptom | 14 days, 28 days
  Reduction of Patient Assessment of Constipation-Symptom (PAC-SYM) questionnaire, a 12-item questionnaire divided into three symptom subscales: abdominal (four items), rectal (three items) and stool (five items). Each item is scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A score reduction represents an improvement of constipation symptoms.
Change in Stool consistency | through study completion, an average of 1 month
  Change in the stool consistency assessed through the 7-point Bristol Stool Form Scale (type 1, type 2, type 3, type 4, type 5, type 6, type 7).
Change of strain evacuation | through study completion, an average of 1 month
  Reduction of number of evacuation with strain
Rescue medication | through study completion, an average of 1 month
  Number of patients who used the rescue medication, nunmber of rescue medication consumed and frequency of use
Change of Quality of Life (QoL) | 14 days, 28 days
  Improvement of QoL through Gastrointestinal Quality of Life Index questionnaire (GIQLI). GiQLI is a 36-item questionnaire, Each item is scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'all the time', 1 = 'most of the time', 2 = 'now and then', 3 = 'rarely' and 4 = 'never'). A score increase represents an improvement of QoL.
Incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, incidence of patients dropped outs. | through study completion, an average of 1 month
  Incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, incidence of patients dropped outs.
Change of strain evacuation | through study completion, an average of 1 month
  Time to event (cox ratio), defined as the first week during which more than 50% of evacuations occurred without strain.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Campus Biomedico, Rome, Lazio
  - IRCCS Istituto Clinico Humanitas, Milan, Lombardy